CLINICAL TRIAL: NCT00347854
Title: Fluorophotometry Evaluation of Lubricant Eye Drops FID 105783
Brief Title: Fluorophotometry Evaluation of Lubricant Eye Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: C-05-06
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Normal, healthy eyes (other than correction for visual acuity)
MeSH Terms: interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- FID 105783 (Experimental)
  Interventions: Other: Systane Free lubricant eye drops
- Visine (Active Comparator)
  Interventions: Other: Visine Tears Lubricant Eye Drops
- Refresh Liquigel (Active Comparator)
  Interventions: Other: Refresh Liquigel Lubricant Eye Drops
- Refresh Plus (Active Comparator)
  Interventions: Other: Refresh Plus Lubricant Eye Drops

INTERVENTIONS:
Other: Systane Free lubricant eye drops
  Arms: FID 105783
Other: Visine Tears Lubricant Eye Drops
  Arms: Visine
Other: Refresh Liquigel Lubricant Eye Drops
  Arms: Refresh Liquigel
Other: Refresh Plus Lubricant Eye Drops
  Arms: Refresh Plus

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of exaggerated use of Lubricant Eye Drops in a population of normal subjects by measuring corneal epithelial permeability to fluorescein.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and over

Exclusion Criteria:

* No sodium fluorescein corneal staining at Screening Visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Epithelial permeability to fluorescein

SECONDARY OUTCOMES:
tear turnover rate

CONTACTS AND LOCATIONS:
Overall Officials: Mike Christensen, Study Director — Alcon Research
Locations (1):
- Alcon, Fort Worth, Texas, United States

REFERENCES:
- [Result] http://www.aaopt.org/evaluation-new-preservation-system-corneal-barrier-function